CLINICAL TRIAL: NCT06591013
Title: Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: the Role of Selection of the Bai Nationality as Donor Source in Terms of Treatment Efficacy and Mechanisms
Brief Title: Efficacy and Mechanism of Fecal Microbiota Transplantation of the Bai Nationality in the Treatment of IBD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yinglei Miao, Director, First Affiliated Hospital of Kunming Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-IBD-240710
Record Dates: First submitted 2024-07-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: fecal microbiota transplantation（FMT）; the Bai Nationality of Yunnan; Intestinal flora; colonoscope; transendoscopic enteral tubing（TET）; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Bai nationality-UC (Experimental): Ulcerative colitis subjects will be treated with bacterial solution from the Bai nationality by colonoscope
  Interventions: Procedure: Fecal microbiota transplantation
- the Han nationality-UC (Experimental): Ulcerative colitis subjects will be treated with bacterial solution from the Han nationality by colonoscope
  Interventions: Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Transplantation of fresh fecal bacterial fluid into the ileocecum of patients with ulcerative colitis via the colonoscopic route

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic, recurrent, non-specific intestinal disease, including ulcerative colitis (UC) and Crohn's disease (CD). Although biological therapy significantly improved the effect of the treatment of ulcerative colitis, but nearly two-thirds of the patient's response to drug treatment. Therefore, new treatments targeting the underlying pathophysiology of UC are critical. Given that alterations in the gut microbiome are strongly associated with disease activity in IBD, many studies have proposed microbiotoy-based therapies, in particular, Fecal microbiota transplantation (FMT) in the treatment of UC. Donor-to-donor variation in treatment with fecal microbiota transplantation may alter treatment efficacy. Therefore, screening high-quality donors can improve efficacy and minimize the risk of adverse effects.

DETAILED DESCRIPTION:
Ulcerative colitis with the changes in the gut microbiota and biodiversity decrease and the change of the relative abundance of advantage bacterium group, a significant reduction in UC patients with intestinal flora diversity, at the species level, thick wall bacteria door bacteria (e.g., clostridium tender) ratio decreases, actinomyces door, the door deformation bacteria such as e. coli), enterobacteriaceae, streptococcus, bacteroides ratio increased.A previous study by team of the investigators found that there were ethnic and regional differences in the incidence of IBD in Yunnan Province, and the incidence of Dai, Bai and Miao was lower than that of Han. Then the related factors were analyzed, among which, the ethnic characteristic diet of Yunnan ethnic minorities can improve the diversity of intestinal flora and viruses, increase the content of probiotics, and is a protective factor for the low incidence of UC.Based on this, donor-to-donor variation in the treatment of fecal microbiota transplantation may alter the therapeutic effect. Therefore, screening high-quality donors can improve efficacy and minimize the risk of adverse effects.Based on this, the investigators asked scientific questions: FMT in the treatment of IBD: the Bai nationality of Yunnan province may be a high quality donor.Our study is aims to FMT in the treatment of IBD, the role of selection of the Bai nationality as donor source in terms of treatment efficacy and mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years inclusive (no limit on gender)
* Confirmed diagnosis of ulcerative colitis for > 3 months, according to established clinical,endoscopic and histologic criteria
* Currently active mild-moderate ulcerative colitis, as measured by a Mayo score of 4-10, in which endoscopy sub-score ≥ 1 and physician's global assessment sub-score ≤ 2
* Written informed consent obtained.

Exclusion Criteria:

* Subjects who are unable to give consent or who have conditions rendering them incapable to answer questionnaires or provide samples.
* Females who are pregnant or actively trying to fall pregnant
* Subjects unwilling to practice an effective method of contraception throughout the study period
* Subjects defined as in remission by the investigator
* Evidence or history of toxic megacolon
* Isolated proctitis < 5 cm
* A diagnosis of Crohn's Disease or indeterminate colitis
* Subjects with perianal disease (e.g. fistulae, pre-existing fissures)
* Significant gastrointestinal surgery e.g. colon resection, colectomy :Minor gastrointestinal surgery will be reviewed on a case by case basis by the investigator;Regarding appendicectomy, only exclude patients who had appendicectomy < 3 months ago)
* Subjects taking antimicrobials (antibiotics, antifungals, antivirals) for any reason, including antibiotics for ulcerative colitis, in the preceding 4 weeks
* Subjects who are steroid dependent and requiring > 20mg prednisone or > 9mg budesonide daily at the time of enrolment
* Subjects who have recently taken or are actively taking or expected to require prohibited medication/s during the study period including follow-up. These include:Rectal therapy including corticosteroid, 5-aminosalicylate within 2 weeks before first FMT;Treatment with biologic agents e.g. infliximab, adalimumab, vedolizumab, within 12 weeks before first FMT;Treatment with other major immunosuppressant agents including calcineurin inhibitors, anti-neoplastic agents, lymphocyte depleting biological agents within 12 weeks before first FMT;Probiotic therapy within 4 weeks before first FMT;Experimental / trial drug protocol involvement within 12 weeks before first FMT;Anti-mycobacterial (TB or MAC) therapy within 4 weeks before first FMT

Allowed concomitant medications:

The following drugs are allowed as long as the dose is stable preceding first FMT for the noted time:

* oral 5-aminosalicylates (stable dose for 4 weeks)
* thiopurines and methotrexate (on medication for ≥ 90 days and dose stable for 4 weeks)
* oral prednisolone (dose ≤ 20mg daily and stable for 2 weeks) During the study, subjects should remained on the same dose of oral 5-aminosalicylate, thiopurine, and methotrexate. For oral prednisolone, dose must be tapered at a rate up to 2.5mg per week so that subjects would be steroid-free by week 8.

Prohibited medications:

The following drugs for are prohibited for the noted time:

* Rectal therapies including corticosteroid, 5-aminosalicylate (for 2 weeks before first FMT and during study period)
* Antibiotics, antibiotics, antifungals, antivirals, probiotic or prebiotic preparations (for 4 weeks before first FMT and during study period)
* Rectal therapies including corticosteroid, 5-aminosalicylate (for 2 weeks before first FMT and during study period)
* Biological therapies or calcineurin inhibitors (for 12 weeks before first FMT and during study period)

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
endoscopic remission or response | 8 to 12 weeks after fecal microbiota transplantation
  a total Mayo score of ≤2 points with no individual sub-score >1 point, and at least a 1 point reduction from baseline in the endoscopy sub-score

SECONDARY OUTCOMES:
Steroid-free clinical remission | 8 to 12 weeks after fecal microbiota transplantation
  combined Mayo sub-scores of 1 or less for rectal bleeding plus stool frequency
Steroid-free clinical response | 8 to 12 weeks after fecal microbiota transplantation
  either a decrease of 3 points or more on the Mayo score, a 50% or greater reduction from baseline in combined rectal bleeding plus stool frequency Mayo sub-scores, or both
Steroid-free endoscopic response | 8 to 12 weeks after fecal microbiota transplantation
  a Mayo endoscopy sub-score of 1 or less, with a reduction of at least 1 point from baseline
Changes in microbial | 0、1、8、12 weeks after fecal microbiota transplantation
  composition,function and metabolite
Difference in microbiome compared between subjects in different treatment arms | 0、1、8、12 weeks after fecal microbiota transplantation
  Difference in microbiome compared between subjects in different treatment arms
Proportion of microbiome derived from recipient, donor or both in subjects who received FMT | 0、1、8、12 weeks after fecal microbiota transplantation
  Proportion of microbiome derived from recipient, donor or both in subjects who received FMT

CONTACTS AND LOCATIONS:
Overall Officials: L Y Miao, Doctor, Principal Investigator — First Affiliated Hospital of Kunming Medical University
Locations (1):
- China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT06591013/Prot_SAP_ICF_000.pdf